CLINICAL TRIAL: NCT06970093
Title: One Anastomosis Gastric Bypass (OAGB) vs Duodeno-jejunostomy For Treatment of Superior Mesenteric Artery Syndrome: A Prospective Randomized Control Trial
Brief Title: Comparison of One Anastomisis Gastric Bypass and Duodeno-Jejunostomy for Treating SMA Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/2024
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Superior Mesenteric Artery Syndrome; Duodenal Obstruction; Weight Loss; Gastrointestinal Disease
Keywords: Superior Mesenteric Artery Syndrome; SMAS; OAGB; One Anastomisis Gastric Bypass; Duodenojejunostomy; Gastrc Bypass; Intestinal Obstruction; Malnutrition; Minimally invasive surgery; Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Superior Mesenteric Artery Syndrome; Duodenal Obstruction; Weight Loss; Gastrointestinal Diseases; Intestinal Obstruction; Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to undergo either One Anastomosis Gastric Bypass (OAGB) or Duodenojejunostomy (DJ).
  Each participant receives one type of surgery, and outcomes are assessed after 12 months of follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OAGB Surgery Group (Experimental): Participants in this arm will undergo One Anastomosis Gastric Bypass (OAGB). The procedure involves creating a long gastric pouch and connecting it to a loop of the jejunum. This reroutes food to bypass the compressed duodenum, aiming to relieve symptoms of Superior Mesenteric Artery Syndrome (SMAS) while preserving nutritional status.
  Interventions: Procedure: One Anastomosis Gastric Bypass
- Duodenojejunostomy Group (Active Comparator): Participants in this arm will undergo Duodenojejunostomy (DJ), a surgical procedure in which a bypass connection is made between the duodenum and the jejunum. This relieves the duodenal compression caused by SMAS and restores normal food passage.
  Interventions: Procedure: Duodenojejunostomy

INTERVENTIONS:
Procedure: One Anastomosis Gastric Bypass — Participants will undergo One Anastomosis Gastric Bypass (OAGB), a laparoscopic bariatric procedure that creates a long narrow gastric pouch and anastomoses it to a loop of jejunum approximately 150-200 cm from the ligament of Treitz. This bypasses the compressed duodenum to relieve symptoms of SMAS while promoting weight gain or nutritional restoration in undernourished patients.
  Other Names: Mini Gastric Bypass
  Arms: OAGB Surgery Group
Procedure: Duodenojejunostomy — Participants will undergo Duodenojejunostomy (DJ), a standard surgical procedure to bypass the compressed segment of the duodenum. It involves creating an anastomosis between the duodenum and the jejunum distal to the point of compression, allowing normal food passage and relieving symptoms of Superior Mesenteric Artery Syndrome.
  Other Names: Duodenal Bypass
  Arms: Duodenojejunostomy Group

SUMMARY:
The goal of this clinical trial is to find out which surgery works better to treat people with a rare condition called Superior Mesenteric Artery Syndrome (SMAS). This condition causes the duodenum to be squeezed between two arteries, leading to severe nausea, vomiting, and weight loss. The researchers are comparing two types of surgery:

* One Anastomosis Gastric Bypass (OAGB)
* Duodeno-jejunostomy (DJ)

The main questions this study will answer are:

* Which surgery improves symptoms and nutritional status better?
* Which surgery leads to fewer complications and better quality of life?

Participants will:

* Be randomly assigned to one of the two surgeries
* Be followed for 12 months after the operation
* Complete follow-up visits and nutritional assessments
* Answer questions about their symptoms and overall well-being

DETAILED DESCRIPTION:
Superior Mesenteric Artery Syndrome (SMAS) is a rare but serious condition where part of the small intestine (the duodenum) gets compressed between major blood vessels. This can cause severe digestive symptoms and weight loss. Surgery is often needed when other treatments do not work.

This prospective randomized controlled trial compares two surgical options to relieve the compression: One Anastomosis Gastric Bypass (OAGB) and Duodeno-jejunostomy (DJ). Both surgeries aim to improve food passage and relieve symptoms, but they work differently and have different effects on digestion and nutrition.

Participants will be randomly assigned to one of the two surgical procedures. The study will collect data before and after surgery on symptoms, nutritional status, complications, and quality of life. Follow-up will continue for 12 months.

The goal is to help surgeons and patients choose the most effective and safest surgical treatment for SMAS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Superior Mesenteric Artery Syndrome (SMAS) based on symptoms and radiologic findings
* No prior gastric or intestinal surgery
* Willingness and ability to participate in follow-up for 12 months

Exclusion Criteria:

* Presence of other gastrointestinal pathologies mimicking SMAS
* Severe comorbidities contraindicating surgery (e.g., advanced cardiac or pulmonary disease)
* History of previous bariatric or upper GI surgery
* Refusal or inability to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Postprandial Symptoms Scores | 12 months
  Change in severity of postprandial symptoms (e.g., nausea, vomiting, early satiety, abdominal pain), assessed using standardized scoring tools: the Numeric Rating Scale (NRS) and the Visual Analog Scale (VAS).
  Both scales range from 0 to 10, where 0 indicates no symptoms and 10 indicates the most severe symptoms imaginable. Higher scores reflect worse symptom severity. The Functional Living Index-Emesis (FLIE) score used to assess nausea and vomiting improvement.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | 12 months
  Change in BMI from baseline to 12 months postoperatively, used to assess nutritional recovery and weight regain after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohey R Elbanna, MD, Study Director — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures will be available to researchers upon reasonable request after the study is published. Data sharing will be considered for academic and clinical research purposes.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 3 months after publication of the primary results and for up to 3 years after publication
Access Criteria: De-identified individual participant data (IPD) and supporting documents such as the study protocol and statistical analysis plan will be available to qualified researchers, academic institutions, or healthcare professionals. These individuals must submit a written request with a sound scientific rationale for secondary analysis. Access will be granted at the discretion of the principal investigator. Approved users must sign a data use agreement to ensure confidentiality and appropriate use. All requests should be sent to the principal investigator's official institutional email address.

REFERENCES:
- [Background] Aleman R, Lo Menzo E, Szomstein S, Rosenthal RJ. Efficiency and risks of one-anastomosis gastric bypass. Ann Transl Med. 2020 Mar;8(Suppl 1):S7. doi: 10.21037/atm.2020.02.03. PMID 32309411
- [Background] Merrett ND, Wilson RB, Cosman P, Biankin AV. Superior mesenteric artery syndrome: diagnosis and treatment strategies. J Gastrointest Surg. 2009 Feb;13(2):287-92. doi: 10.1007/s11605-008-0695-4. Epub 2008 Sep 23. PMID 18810558
- [Background] Zaraket V, Deeb L. Wilkie's Syndrome or Superior Mesenteric Artery Syndrome: Fact or Fantasy? Case Rep Gastroenterol. 2015 Jun 5;9(2):194-9. doi: 10.1159/000431307. eCollection 2015 May-Aug. PMID 26120301
- [Background] Lee TH, Lee JS, Jo Y, Park KS, Cheon JH, Kim YS, Jang JY, Kang YW. Superior mesenteric artery syndrome: where do we stand today? J Gastrointest Surg. 2012 Dec;16(12):2203-11. doi: 10.1007/s11605-012-2049-5. Epub 2012 Oct 18. PMID 23076975
- [Background] Welsch T, Buchler MW, Kienle P. Recalling superior mesenteric artery syndrome. Dig Surg. 2007;24(3):149-56. doi: 10.1159/000102097. Epub 2007 Apr 27. PMID 17476104